CLINICAL TRIAL: NCT06862206
Title: A Multicentre, Single Arm, Non-interventional, Prospective Study to Assess Demographic Characteristics and Patient Reported Outcomes in Patients With Severe Eosinophilic Asthma Treated With Benralizumab in China
Brief Title: This is a Non-interventional, Study to Assess Demographic Characteristics and Patient Reported Outcomes in China Patients With SEA Treated With Benralizumab
Acronym: SPEED
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00131
Record Dates: First submitted 2025-03-03; First posted 2025-03-06 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — benralizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- benralizumab group: non-interventional
  Interventions: Other: benralizumab

INTERVENTIONS:
Other: benralizumab — non-interventional

SUMMARY:
The objective of this study is to collect empirical data that elucidates the clinical profile and therapeutic efficacy of benralizumab among the patients aged 12 years and above, with severe eosinophilic asthma. The study will focus on the early treatment response, treatment outcomes and the change in asthma control of benralizumab therapy in a real-world setting in China. This study will also describe the physician-reported reasons for discontinuation and switching of benralizumab therapy.

ELIGIBILITY:
Inclusion criteria -Patients are eligible to be included in the study only if all of the following criteria apply:

* Patients must to be 12 years old (inclusive) at the time of signing the informed consent.
* Patients with severe eosinophilic asthma prescribed with benralizumab at the discretion of the clinician.
* Blood EOS≥150/ul in the 3 months prior to or EOS≥300/ul in the 1 year prior to the time of signing the informed consent.
* Participating patients and/or their legally authorized representative must provide signed and dated written informed consent form prior to any study specific procedures.

Exclusion criteria

-Patients should not enter the study if any of the following exclusion criteria are fulfilled:

* Patients currently participating in any other clinical trial.
* Known history of allergy or reaction to any component of the study treatment formulation.
* Malignancy of any kind.
* Patients with prior or ongoing treatment with benralizumab.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: severe eosinophilic asthma
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
asthma control questionnaire | Week 8
  To describe the change in asthma control questionnaire at early time point after initiation of benralizumab

SECONDARY OUTCOMES:
asthma control questionnaire | week 1, 2, 4, 8, 16, 24, 40 and 56.
  * Changes from baseline in ACQ-6 at week 1, 2, 4, 16, 24, 40 and 56 after initiation of benralizumab.
  * The percentage of patients well controlled (defined as ACQ-6 score ≤0.75), partially controlled (defined as ACQ-6 score >0.75 and < 1.5) and uncontrolled (defined as ACQ-6 score ≥1.5) at week 1, 2, 4, 8, 16, 24, 40 and 56.
  * The percentage of patients who had clinically meaningful change of ACQ-6 (defined as at least (≥) 0.5-unit improvement in ACQ-6 score) at the end of treatment at week 1, 2, 4, 8, 16, 24, 40 and 56.
changes in lung function | week 8, 16 and 56
  Changes from baseline in pre-BD FEV1 at week 8, 16 and 56 after initiation of benralizumab.

CONTACTS AND LOCATIONS:
Overall Officials: chen wang, PhD, Principal Investigator — China-Japan Friendship Hospital
Locations (16):
- China (16):
  - Research Site, Beijing
  - Research Site, Binzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Huzhou
  - Research Site, Jinan
  - Research Site, Jinhua
  - Research Site, Jining
  - Research Site, Linyi
  - Research Site, Mianyang
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Shanxi
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/